CLINICAL TRIAL: NCT06730360
Title: Clinical and Radiographic Assessment of Photobiomodulated MTA Pulpotomy in Immature First Permanent Molars with Irreversible Pulpitis: a Randomized Controlled Clinical Trial
Brief Title: Clinical and Radiographic Assessment of Photobiomodulated MTA Pulpotomy in Immature First Permanent Molars with Irreversible Pulpitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Peter Samir, assistant lecturer, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A0109024PP
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-09

CONDITIONS: Dental Caries; Irreversible Pulpitis
Keywords: Irreversible pulpitis; Immature permanent molars; Vital pulp therapy (VPT); Mineral trioxide aggregate (MTA); Photobiomodulation (PBM)
MeSH Terms: conditions — Dental Caries | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MTA Pulpotomy without Photobiomodulation (Active Comparator): Participants will receive MTA (Mineral Trioxide Aggregate) pulpotomy as a standard treatment without the application of photobiomodulation (low-level laser therapy).
  Interventions: Procedure: MTA Pulpotomy without photobiomodulation
- MTA Pulpotomy with Photobiomodulation (Experimental): Participants will receive MTA (Mineral Trioxide Aggregate) pulpotomy treatment enhanced with photobiomodulation (low-level laser therapy). The laser will be applied to pulp stumps before the placement of MTA to promote healing and reduce inflammation.
  These entries should resolve the error and align with your protocol.
  Interventions: Procedure: MTA Pulpotomy with Photobiomodulation (LLLT)

INTERVENTIONS:
Procedure: MTA Pulpotomy without photobiomodulation — This intervention involves the application of Mineral Trioxide Aggregate (MTA) to the pulp chamber after the removal of the coronal pulp tissue in first permanent molars with irreversible pulpitis. The procedure is performed without the use of photobiomodulation (low-level laser therapy). The MTA is placed as a seal to preserve the vitality of the remaining radicular pulp.
  Arms: MTA Pulpotomy without Photobiomodulation
Procedure: MTA Pulpotomy with Photobiomodulation (LLLT) — This intervention combines MTA pulpotomy with photobiomodulation (low-level laser therapy). After performing the MTA pulpotomy, low-level laser therapy is applied to the pulp stumps to reduce inflammation, promote healing, and modulate pain. The laser therapy uses specific wavelengths of light to stimulate cellular activity and enhance the regeneration of pulp tissue.
  Arms: MTA Pulpotomy with Photobiomodulation

SUMMARY:
This study evaluates the effectiveness of photobiomodulation (PBM) in conjunction with mineral trioxide aggregate (MTA) pulpotomy for treating irreversible pulpitis in immature first permanent molars. PBM, also known as low-level laser therapy (LLLT), is used to enhance healing, reduce inflammation, and manage pain in young teeth. The randomized clinical trial involves 72 children aged 6-9 years, divided into two groups: one receiving MTA pulpotomy alone and the other receiving MTA pulpotomy with PBM. Clinical and radiographic outcomes will be assessed at intervals over 15 months. This research aims to determine the combined therapy's efficacy in improving pulp healing and reducing post-operative discomfort compared to MTA alone.

DETAILED DESCRIPTION:
This randomized controlled trial evaluates the clinical and radiographic outcomes of MTA pulpotomy, with and without PBM, for immature permanent molars diagnosed with irreversible pulpitis. The study includes two parallel groups of 36 children each. Group I will undergo MTA pulpotomy alone, while Group II will receive PBM treatment alongside MTA pulpotomy.

PBM employs low-level laser therapy to stimulate pulp tissue regeneration, enhance mitochondrial activity, and reduce inflammation and pain, thereby potentially improving MTA pulpotomy outcomes. Key inclusion criteria involve children with deep carious lesions and clinical signs of irreversible pulpitis but without pulpal necrosis. Follow-up will occur at 3, 6, 12, and 15 months post-treatment to evaluate success based on the absence of clinical symptoms (e.g., pain, tenderness) and radiographic indicators of healing.

By comparing these two approaches, the study aims to provide insights into PBM's role as an adjunctive therapy for vital pulp preservation, particularly in pediatric dentistry.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6 to 9 years.
* Non-contributory medical history (healthy otherwise).
* Presence of carious first permanent molars with the following characteristics:
* Deep caries extending to ≥2/3 of dentin.
* Positive response to cold testing.
* Clinical diagnosis of irreversible pulpitis (moderate or severe), with or without periapical periodontitis.
* Restorable tooth.
* Probing pocket depth and mobility within normal limits.
* No signs of pulpal necrosis, including sinus tract or swelling.

Exclusion Criteria:

* Insufficient bleeding after pulp exposure (indicating necrotic or partially necrotic pulp).
* Presence of systemic or medical conditions that may contraindicate participation.
* Teeth with unrestorable structure.
* Teeth showing signs of pulpal necrosis, such as the presence of a sinus tract or swelling.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2024-10-10 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
Clinical Success of Pulpotomy Treatment | 15 months post-treatment (assessed at 3, 6, 12, and 15 months).
  Evaluation of clinical signs and symptoms (absence of pain, tenderness to percussion, sinus tract, or swelling). Treatment is considered successful if these are absent at all follow-up visits.

SECONDARY OUTCOMES:
Radiographic Healing | 15 months post-treatment (assessed at 6, 12, and 15 months).
  Assessment of radiographic evidence of healing, including no periapical rarefaction, root resorption, or new furcal pathosis. Success is determined by achieving a PAI (Periapical Index) score of 1 or 2, or reduction in PAI score if preoperative rarefaction is present.
  Periapical Index (PAI) Scale: 1 to 5
  Interpretation:
  1: Normal periapical structures (better outcome) 5: Severe changes with evident bone destruction (worse outcome).
Root Development Progression | 15 months post-treatment (assessed at 6, 12, and 15 months)
  Radiographic evaluation of root maturity and the formation of a hard tissue bridge

OTHER OUTCOMES:
Postoperative Pain Intensity | 2 days post-treatment.
  Measured using the Wong-Baker Faces Pain Rating Scale to assess postoperative pain levels.
  Wong-Baker Facial Pain Rating Scale Scale: 0 to 10
  Interpretation:
  0: No pain (better outcome) 10: Worst pain imaginable (worse outcome).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided